CLINICAL TRIAL: NCT02175953
Title: Psychotherapeutical Short-term Intervention for Caregivers of Persons With Dementia
Brief Title: Short-term Caregiver Psychotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rostock (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Ingo Kilimann, Neurologist, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RO020
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Caregiver Burden of People With Dementia
Keywords: caregiver burden; stress; depression; dementia
MeSH Terms: conditions — Caregiver Burden; Depression; Dementia | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventiongroup (Experimental): Psychotherapy
  Interventions: Behavioral: Psychotherapy
- Waitling list group (No Intervention): waiting list

INTERVENTIONS:
Behavioral: Psychotherapy — The program is designed for 10 participants and consists of two modules of caregiver education followed by ten psychotherapeutic group modules. The major overarching topics will be (i) caregiver´s emotional and physical limits, (ii) conscious and unconscious feelings and emotions towards the people with dementia and (iii) activation of caregivers´ social resources. Duration of each module is planned to be 90 minutes including a relaxation exercise at the end of each module.
  Arms: Interventiongroup

SUMMARY:
This study is to test the feasibility (pilot part) and efficacy (phase IIa part) of a specifically on the needs of caregivers of people with dementia composed new short-term psychotherapeutical intervention.

DETAILED DESCRIPTION:
This prospective study will be offered to caregivers from the out patient clinic of the Department of Psychosomatic Medicine of the University Rostock Medical Center. In a first pilot study with 10 participants without control group, we tested the feasability and acceptance of the program (completed 2/2015). From 4/2015 a phase IIa study started with 10 participants in the intervention group and 10 in the control groups (will be organized by waiting list). The program consists of two modules of caregiver education followed by ten psychotherapeutic group modules. Duration of each module is planned to be 90 minutes including a relaxation exercise at the end of each module. Primary outcomes are the feasibility, acceptance and the effect on caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* caregiver of a person with dementia
* willing to participate in all 12 modules of the program

Exclusion Criteria:

* current psychotherapy or antidepressive medication for less than 6 month
* major depression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in perceived self-efficacy directly and 3 month after psychotherapeutical intervention and reduction of symptoms of depression | before intervention, 0 and 3 month after end of intervention
  SWE, a german self-efficacy self-rating scale, will be used for self-efficacy measurement AND ADS (German Version of the CES-D Scale) for measurement for symptoms of depression

SECONDARY OUTCOMES:
reduction of perceived burden of care | before intervention, 0 and 3 month after end of intervention
  We will be using the Zarit-Burden-Interview to measure the perceived burden of care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK.
- [Background] Weissman MM, Sholomskas D, Pottenger M, Prusoff BA, Locke BZ. Assessing depressive symptoms in five psychiatric populations: a validation study. Am J Epidemiol. 1977 Sep;106(3):203-14. doi: 10.1093/oxfordjournals.aje.a112455. PMID 900119